CLINICAL TRIAL: NCT05303233
Title: Analgesic Efficacy of IPACK Versus Selective Tibial Nerve Block in Patients Scheduled for Anterior Cruciate Ligament Reconstruction Under General Anaesthesia With an Adductor Canal Block: a Randomized Controlled Double-blinded Trial
Brief Title: IPACK or Selective Tibial Nerve Block for ACL Reconstruction With an Adductor Canal Block
Acronym: TIPACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Prof. Dr. med. Eric Albrecht, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CER-VD 2021-02474
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Analgesia
Keywords: Regional anesthesia; Selective tibial nerve block; IPACK; Anterior cruciate ligament reconstruction; Multimodal analgesia; Local anesthetics
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TIBIAL group (Experimental): All patients allocated to the TIBIAL group will receive an adductor canal block with 20ml of ropivacaine 0.75% and a selective tibial nerve block with 5 ml of ropivacaine 0.75% prior to surgery,
  Interventions: Procedure: Selective tibial nerve block
- IPACK group (Active Comparator): All patients allocated to the IPACK group will receive an adductor canal block with 20ml of ropivacaine 0.75% and an IPACK with 20ml of ropivacaine 0.2% prior to surgery.
  Interventions: Procedure: IPACK

INTERVENTIONS:
Procedure: Selective tibial nerve block — The selective tibial nerve block will be performed on the popliteal crease following sterilization of the area. The probe will be placed in a transverse position at the popliteal crease to visualize the popliteal artery and the tibial nerve in short axis. A 21-gauge 50mm insulated facet tip needle (SonoPlex® STIM, Pajunk, Geisingen, DE) will be inserted in-plane with the ultrasound bean from a medial to lateral direction. Once the needle tip is adjacent to the tibial nerve, 5 ml of ropivacaine 0.75% will be injected to achieve an adequate spread of local anaesthetics around the nerve.
  Arms: TIBIAL group
Procedure: IPACK — The IPACK will be performed on the popliteal crease following sterilization of the area. The probe will be placed in a transverse position proximal to the popliteal crease to visualize the popliteal artery in short axis. A 21-gauge 100 mm insulated facet tip needle (SonoPlex® STIM, Pajunk, Geisingen, DE) will be inserted in-plane with the ultrasound beam, in a lateral to medial direction, between the popliteal artery and the posterior capsule, where twenty mL of ropivacaine 0.2% will be injected under ultrasound guidance. The distribution of local anaesthetics will be observed above the posterior capsule.
  Arms: IPACK group

SUMMARY:
The purpose of this study is to compare the analgesic efficacy of the combination of an adductor canal and selective tibial nerve blocks versus adductor canal block and IPACK after ACL reconstruction under general anaesthesia.

DETAILED DESCRIPTION:
The hypothesis of this study is that a combined adductor canal and selective tibial nerve block provides better analgesia than a combined adductor canal block and IPACK in patients undergoing anterior cruciate ligament reconstruction.

This randomized controlled trial will include two groups: an adductor canal block plus IPACK group (group IPACK) and an adductor canal block plus tibial selective nerve block group (group TIBIAL). After written informed consent, patients will be allocated to one of the groups, following a computer-generated list of randomization.

Prior to surgery, all patients will have an adductor canal block with 20ml of ropivacaine 0.75%. In group TIBIAL the patient will receive in addition a selective tibial nerve block with 5 ml of ropivacaine 0.75%. In group IPACK the patient will receive in addition an IPACK with 20ml of ropivacaine 0.2%. In both groups, patients will have the surgery under general anaesthesia with a multimodal analgesic regimen inclusive of iv dexamethasone 8 mg, iv magnesium sulfate 40 mg.kg-1, iv ketorolac 30 mg, and iv acetaminophen 1000 mg.

After surgery, all patients will be prescribed an iv patient-controlled analgesia (PCA) of morphine (boluses of 2 mg available every 10 min, maximum of 40 mg every 4 hours) along with oral acetaminophen (1000 mg every 6 h) and oral ibuprofen (400 mg every 8 hours). Oral ondansetron 4 mg every 8 hours will be available on request in case of nausea or vomiting.

The primary outcome will be the cumulative iv morphine consumption at 24 h postoperatively. Secondary outcomes will include pain- and functional-related outcomes. Pain-related outcomes include cumulative morphine consumption at 2h and 48h postoperatively, rest and dynamic pain scores and rate of PONV at 2 h, 24 h and 48 h postoperatively. Early functional-related outcomes include range of motion, strength and walking distance at 24 h and 48 h postoperatively. Late functional-related outcomes include range of motion, strength, hop distance, agility test, Y balance test, Anterior Cruciate Ligament Return to Sport After Injury Scale (ACL-RSI) and International Knee Documentation Committee Scale (IKDC) at 4 and 8 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA score I-III
* 18 years or older
* Scheduled for elective primary ACL reconstruction
* Signature of consent form

Exclusion Criteria:

* Refusal or inability for informed consent
* Known allergies to ropivacaine, acetaminophen, ibuprofen, ketorolac, morphine, sufentanyl, ondansetron or dexamethason
* Secondary surgical revision
* Opioid treatment such as morphine, hydrocodone, hydromorphone, tramadol, methadone, fentanyl, buprenorphine or codeine
* Bleeding diathesis
* Neurological deficit
* Known renal insufficiency (eGFR <45 ml/min)
* Known hepatic insufficiency (Child score B or C)
* Pregnancy or lactating
* Alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Total intravenous morphine consumption | 1 day postoperatively
  Consumption in mg

SECONDARY OUTCOMES:
Total intravenous morphine consumption | 2 hours and 2 days postoperatively
  Consumption in mg
Resting and dynamic pain score | 2 hours, 1 day and 2 days postoperatively
  Numeric Rating Scale (NRS), 0-10 where 0 is no pain and 10 is the worst pain imaginable
Incidence of postoperative nausea and vomiting | 2 hours, 1 day and 2 days postoperatively
  Presence of nausea and vomiting in the postoperative period
Range of motion | 1 day and 2 days postoperatively
  Joint motion in degrees
Quadriceps strength | 1 day and 2 days postoperatively
  Ordinal scale of 1-5, with 5 being the maximal developed strength compared with the opposite side
Walking distance | 1 day and 2 days postoperatively
  Distance in meters
Range of motion | 4 months and 8 months postoperatively
  Joint motion in degrees
Concentric quadriceps strength and concentric hamstring strength | 4 months and 8 months postoperatively
  Percentage of strength as compared with the opposite leg
Single hop distance, triple hop distance and crossover triple hop distance | 4 months and 8 months postoperatively
  Percentage of distance as compared with the opposite leg
Agility test | 4 months and 8 months postoperatively
  Time in second
Y balance test | 4 months and 8 months postoperatively
  Distance in cm
Anterior Cruciate Ligament Return to Sport After Injury Scale score | 4 months and 8 months postoperatively
  Score in percentage
International Knee Documentation Committee Scale score | 4 months and 8 months postoperatively
  Score in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Eric Albrecht, M.D., Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- University Hospital of Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chuaychoosakoon C, Parinyakhup W, Wiwatboworn A, Purngpiputtrakul P, Wanasitchaiwat P, Boonriong T. Comparing post-operative pain between single bundle and double bundle anterior cruciate ligament reconstruction: a retrospective study. BMC Musculoskelet Disord. 2021 Sep 3;22(1):753. doi: 10.1186/s12891-021-04635-5. PMID 34479511
- [Background] Smith JH, Belk JW, Kraeutler MJ, Houck DA, Scillia AJ, McCarty EC. Adductor Canal Versus Femoral Nerve Block after Anterior Cruciate Ligament Reconstruction: A Systematic Review of Level I Randomized Controlled Trials Comparing Early Postoperative Pain, Opioid Requirements, and Quadriceps Strength. Arthroscopy. 2020 Jul;36(7):1973-1980. doi: 10.1016/j.arthro.2020.03.040. Epub 2020 Apr 18. PMID 32315764
- [Background] Jansen TK, Miller BE, Arretche N, Pellegrini JE. Will the addition of a sciatic nerve block to a femoral nerve block provide better pain control following anterior cruciate ligament repair surgery? AANA J. 2009 Jun;77(3):213-8. PMID 19645171
- [Background] Silverman ER, Vydyanathan A, Gritsenko K, Shaparin N, Singh N, Downie SA, Kosharskyy B. The Anatomic Relationship of the Tibial Nerve to the Common Peroneal Nerve in the Popliteal Fossa: Implications for Selective Tibial Nerve Block in Total Knee Arthroplasty. Pain Res Manag. 2017;2017:7250181. doi: 10.1155/2017/7250181. Epub 2017 Feb 2. PMID 28260964
- [Background] Stebler K, Martin R, Kirkham KR, Lambert J, De Sede A, Albrecht E. Adductor canal block versus local infiltration analgesia for postoperative pain after anterior cruciate ligament reconstruction: a single centre randomised controlled triple-blinded trial. Br J Anaesth. 2019 Aug;123(2):e343-e349. doi: 10.1016/j.bja.2019.04.053. Epub 2019 May 24. PMID 31130273
- [Background] Martin R, Kirkham KR, Ngo THN, Gonvers E, Lambert J, Albrecht E. Combination of femoral triangle block and infiltration between the popliteal artery and the capsule of the posterior knee (iPACK) versus local infiltration analgesia for analgesia after anterior cruciate ligament reconstruction: a randomized controlled triple-blinded trial. Reg Anesth Pain Med. 2021 Sep;46(9):763-768. doi: 10.1136/rapm-2021-102631. Epub 2021 May 26. PMID 34039734
- [Background] van der Wal M, Lang SA, Yip RW. Transsartorial approach for saphenous nerve block. Can J Anaesth. 1993 Jun;40(6):542-6. doi: 10.1007/BF03009739. PMID 8403121